CLINICAL TRIAL: NCT00936728
Title: White Wine for Appetite Loss: A Randomized, Controlled, Non-Blinded Trial
Brief Title: White Wine or Nutritional Supplement in Improving Appetite in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC08C6; NCI-2009-01130 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA124614 (NIH); RC08C6 (Other: Mayo Clinic Cancer Center); 09-000862 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2009-07-06; First posted 2009-07-10 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (white wine) (Experimental): Patients consume white wine twice daily for 3-4 weeks.
  Interventions: Dietary Supplement: white wine; Other: questionnaire administration
- Arm B (non-wine nutritional supplement) (Active Comparator): Patients receive an oral non-wine nutritional supplement (e.g., Boost or Ensure) twice daily for 3-4 weeks.
  Interventions: Other: therapeutic nutritional supplementation; Other: questionnaire administration

INTERVENTIONS:
Other: therapeutic nutritional supplementation — Given orally
  Arms: Arm B (non-wine nutritional supplement)
Dietary Supplement: white wine — Given orally
  Arms: Arm A (white wine)
Other: questionnaire administration — Ancillary studies

SUMMARY:
RATIONALE: It is not yet know whether white wine is more effective than a nutritional supplement in improving appetite.

PURPOSE: This randomized clinical trial is studying white wine to see how well it works compared with a nutritional supplement in improving appetite in patients with cancer

DETAILED DESCRIPTION:
OBJECTIVES:

I. To compare white wine (Arm A) to non-wine nutritional supplement (Arm B) for the treatment of cancer-associated anorexia.

II. To evaluate the side effect profile of white wine (Arm A).

OUTLINE: Patients are stratified according to primary malignant disease (lung vs gastrointestinal vs other [specify]), severity of weight loss (excluding peri-operative weight loss) within the past 2 months (< 4.6 kg [< 10 lbs] vs >= 4.6 kg [>= 10 lbs]), age (< 50 years vs >= 50 years), and planned concurrent chemotherapy or radiation (yes vs no).

Patients are randomized to 1 of 2 arms.

ARM A: Patients consume white wine with =< 15% alcohol content twice daily for 3-4 weeks.

ARM B: Patients receive an oral non-wine nutritional supplement (e.g., Boost or Ensure) twice daily for 3-4 weeks.

After completion of study treatment, patients are followed up every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Incurable, invasive malignancy
* Able to reliably take the study intervention as prescribed in this protocol
* No prior or current history of alcoholism
* Alert and mentally competent
* Physician estimates that patient has lost >= 5 pounds (2.3 kg) in weight =< 2 months (excluding peri-operative weight loss; documented weight loss not required) and/or have estimated caloric intake of < 20 cal/kg daily (no further documentation necessary other than an affirmative answer to this statement)
* Patient perceives loss of appetite and/or weight as a problem; NOTE: Documentation not necessary
* Concurrent chemotherapy and/or radiotherapy are permitted
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willingness to abstain completely from alcohol for 4 weeks, except as prescribed in this trial; NOTE: Patients assigned to the non-wine nutritional supplement (Arm B) must be willing to abstain from wine and other alcoholic beverages for 3-4 weeks; Patients assigned to the white wine (Arm A) are allowed to take a nutritional supplement, such as Ensure or Boost if they choose to
* Ability to complete questionnaire(s) by themselves or with assistance
* Willingness to return to MCCRC enrolling institution for follow-up
* Patients in whom the use of progestational agents is anticipated are not permitted to be on this study
* Short-term use of dexamethasone around days of intravenous chemotherapy is allowed for protection against emesis, but dexamethasone for appetite stimulation is not permitted

Exclusion Criteria:

* Receiving tube feedings or parenteral nutrition
* Current (=< 1 month) or planned treatment with adrenal corticosteroids (short-term use of dexamethasone around days of chemotherapy is allowed for protection against emesis), androgens, or progestational agents; EXCEPTION: Inhalant, topical, or optical steroid use is permissible
* Progestational agent (such as megestrol acetate) planned to be initiated over the next 30 days; NOTE: Patients who have been on megestrol acetate for > 1 month and are still on it and otherwise meet the eligibility criteria are permitted to enroll on this protocol and remain on megestrol acetate
* Known mechanical obstruction of the alimentary tract, malabsorption, or intractable vomiting (> 5 episodes/week)
* Symptomatic or untreated brain metastases
* Any of the following as this regimen may be harmful to a developing fetus or nursing child: pregnant women, nursing women, and men or women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2009-07 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-04-17 (Actual)

PRIMARY OUTCOMES:
Difference in the percentage of patients who report an improvement in their appetite over the intervention period | First 3 weeks

SECONDARY OUTCOMES:
Differences in the percentage of patients who manifest weight stability, defined as weight gain of at least 5% of baseline | At one month
Overall survival | Every 6 months for 2 years
Incidence of study intervention-related toxicity | Prior to registration and at week 3-4
Patient-reported quality of life (QOL) as measured by the Functional Assessment of Anorexia/Cachexia Therapy (FAACT) appetite scale | Prior to study intervention and then weekly

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, M.D., Study Chair — Mayo Clinic; Tom R. Fitch, M.D., Principal Investigator — Mayo Clinic; Amber L. Isley, M.D., Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Geisinger Medical Center, Danville, Pennsylvania